CLINICAL TRIAL: NCT05767541
Title: Comparative Effects of Pilates Exercises Versus Resistance Exercises on Measures of Physical Functioning Among Geriatric Population With Sarcopenia. a Randomized Clinical Trial
Brief Title: Pilates Exercises Versus Resistance Exercises Among Geriatric Population With Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Syeda Ariba Shoaib, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2642
Record Dates: First submitted 2022-12-24; First posted 2023-03-14 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Resistance training; Exercise Movement Techniques
MeSH Terms: conditions — Sarcopenia | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates group (Experimental): The Pilates technique consists of a series of low-impact exercises that build strength and flexibility throughout the body. All exercises performed 3 days in a week, 3 visits per week total of 9 sessions. In first week participants will perform 1 set of each exercise with 10 repetitions. In second week 2 sets of each exercise with 12 repetitions and in the third week both groups will perform 3 sets of each exercise with 15 repetitions with a rest interval of 2-3 minutes between sets.
  Interventions: Other: Pilates exercises
- Resistance group (Active Comparator): Resistance exercises are anaerobic physical exercises, uses low number of repetitions with adjustable intensity contribute to hypertrophy of the muscle fibers and increase in muscle strength. All exercises performed 3 days in a week, 3 visits per week total of 9 sessions. In first week participants will perform 1 set of each exercise with 10 repetitions. In second week 2 sets of each exercise with 12 repetitions and in the third week both groups will perform 3 sets of each exercise with 15 repetitions with a rest interval of 2-3 minutes between sets.
  Interventions: Other: Resistance exercises

INTERVENTIONS:
Other: Pilates exercises — The Pilates technique consist of hundred, swimming, prone leg lift, single leg stretch, spine stretch forward, arm circles, imprint and release, one leg circles and mini squat.
  Arms: Pilates group
Other: Resistance exercises — Resistance training include leg press, shoulder press, bench press, back arm press, seated row, knee extension, leg curl and seated calf raise
  Arms: Resistance group

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of two exercises to improve physical functioning of older adults with sarcopenia. the primary aim of this RCT is:

To measure the influence of pilates exercises versus resistance training in elderly with sarcopenia.

To introduce an affordable, effective and safe exercise care program, which prioritizes to make geriatric population independent.

Participants will be assessed for all outcome measures change at baseline and after 3 weeks following an exercise intervention. Participants enrolled in pilates exercise group will receive total of 9 exercises and participants enrolled in resistance exercise group will receive total of 8 exercises.

DETAILED DESCRIPTION:
A total sample of 70 of geriatric population with sarcopenia will be collected from Dow University Hospital Ojha. Non-probability purposive sampling technique will be used. Participants will be screened and referred from medicine, family medicine and neurology OPD to physiotherapy OPD. Outcome measure assessment will be performed in all patients at two time points: baseline and follow up at the end of last session.

Outcome measures include short physical performance battery assessment tool (SPPB). Strength and gait are first evaluated by the ability to perform the tasks of getting up and sitting on a chair five consecutive times and performing the walking speed test (3 meters), Time up and go test, sit and reach test, and 2-minute step test as a measure of physical functioning.

After complete assessment at baseline all participants will be randomized to different treatment groups using 70 opaque sealed envelopes containing notes written with "new treatment" or "Standard treatment" on (n= 35 of each). The envelops will be scrambled before each participant allow to draw an envelope and thus find out in which group they will be allocated. Treatment will be provided to both groups. Group 1 will be provided with pilates exercises and group 2 will be provided with resistance exercises. Both groups will perform generalized warm up for up to 10 minutes at the beginning and 10 minutes of relaxation exercises at the end of treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Referred and screened patients with sarcopenia from medicine, family medicine and neurology OPD at Dow University Hospital Ojha Campus, Karachi.
* Patients from 60 to 70 years of age
* Both male and female.
* Patients who consent to participate

Exclusion Criteria:

* Being bedridden
* Implanted pacemaker
* Recent history of any fracture
* Patients with cognitive & neurological impairment
* Already enrolled in any exercise intervention program
* Known case of patients with malignancy
* Patients on steroids

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Short physical performance battery assessment tool. | 3 weeks, change from baseline
  The SPPB assesses physical performance through balance, strength, and gait.
  .Each test is scored from 0 (inability to perform the task) to 4 points (best test performance).The SPPB total score ranges from 0 (worst performance) to 12 points (best performance) and categorically evaluates performance in the tests using three classes of scores: three classes: 0-6 points (poor performance), 7-9 points (moderate performance), and 10-12 points (good performance).

SECONDARY OUTCOMES:
Time up and go test | 3 weeks, change from baseline
  TIME UP AND GO TEST: To evaluate agility and dynamic balance this is essential for tasks that demands quick movements.
sit and reach test | 3 weeks, change from baseline
  SIT AND REACH TEST: It determines the lower back and hamstring flexibility. Which is necessary for proper gait pattern, good posture and multiple movement task.
2-minute step test | 3 weeks, change from baseline
  2-MINUTE STEP TEST: To assess aerobic fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Syeda Ariba Shoaib, Principal Investigator — Dow University of Heath Sciences
Locations (2):
- Pakistan (2):
  - Dow University of Health and Sciences, Karachi, Sindh
  - Dow University of Health and Sciences, Karachi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mueller D, Redkva PE, Fernando de Borba E, Barbosa SC, Krause MP, Gregorio da Silva S. Effect of mat vs. apparatus pilates training on the functional capacity of elderly women. J Bodyw Mov Ther. 2021 Jan;25:80-86. doi: 10.1016/j.jbmt.2020.11.012. Epub 2020 Nov 16. PMID 33714516
- See also: Effect of mat vs. apparatus pilates training on the functional capacity of elderly women — https://pubmed.ncbi.nlm.nih.gov/33714516/